CLINICAL TRIAL: NCT00351429
Title: Evaluating the Safety and Efficacy of Polyglycolic Acid Suture in Ophthalmic Surgical Procedures
Brief Title: Study of PGA Suture in Ophthalmology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: A. Heber, Aurolab
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1010510
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Trabeculectomy; Sutures
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Polyglycolic acid suture

INTERVENTIONS:
Device: Polyglycolic acid suture — PGA suture used in Trabeculectomy surgery
  Other Names: Aurocryl

SUMMARY:
To evaluate the safety and efficacy of polyglycolic acid suture in ophthalmic surgical procedures

DETAILED DESCRIPTION:
The sutures are classified into non-absorbable and absorbable sutures. Violet braided polyglycolic acid suture is the synthetic absorbable suture used in wound closure in ophthalmology, cardiology, neurology and plastic & reconstructive surgeries. In ophthalmology, PGA sutures are used in Trabeculectomy (Glaucoma), Orbit and Oculoplasty, Lid and Socket Reconstruction, Squint, ptosis and retinal detachment surgeries.

Glaucoma patients who met the inclusion criteria were recruited for this study. Uniform surgery and suturing technique was performed in all patients (Trabeculectomy with IOL implantation). Surgeon assessed suture characteristics during surgery and wound integrity at the end of surgery.

Patients were followed up during 1 day, 1 month and 3 months post operatively. Visual acuity, Intraocular Pressure (IOP), suture characteristics, wound integrity, inflammation and conjunctival status were examined during each follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Trabeculectomy with IOL implantation
* Current residence within 60 kms of madurai

Exclusion Criteria:

* Life threatening illness
* Immunosuppressive disorders
* Chronic infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Suture characteristics | 1 month, 3 months

SECONDARY OUTCOMES:
Bleb characteristics | 1 month, 3 months
Conjunctival status | 1 month, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Krishnadas, DO, Dip NB, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India